CLINICAL TRIAL: NCT07165821
Title: Effects of an Interpersonal Communication Skills Training Program on Medication Adherence of Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suranaree University of Technology (Other)
Responsible Party: Principal Investigator, Sakda Khumkom, Sakda Khumkom, Ph.D. , Asst.Prof., School of Psychiatric Nursing, Institue of Nursing, Suranaree University of Technology, Suranaree University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NursingSUT
Record Dates: First submitted 2025-08-24; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Psychosis; Remission; Non-Adherence, Medication
Keywords: Medication Adherence; Schizophrenia; Interpersonal Communication Skills Training
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Medication Adherence

STUDY DESIGN:
Masking Description: Participants who met the inclusion criteria were randomly assigned using a simple lottery method into an experimental group (n = 20) and a control group (n = 20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): The group of patients who received Interpersonal Communication Skills Training Program
  Interventions: Behavioral: Interpersonal Communication Skills Training Program
- Control group (Other): The group of patients who received routine psychiatric nursing care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Interpersonal Communication Skills Training Program — This program was developed based on DeVito's communication theory and integrated with the positive reinforcement-based interpersonal communication training developed by Thiengwiriyakul et al.(11) This program was evaluated by a panel of three experts-a psychiatrist, a psychiatric nurse, and a psychiatric nursing academic-who assessed content relevance, appropriateness, and language clarity. After revisions based on their feedback, the program achieved a Content Validity Index (CVI) of 0.93, exceeding the acceptable threshold.
  Arms: Experiment group
Behavioral: Usual care — Received routine psychiatric nursing care
  Arms: Control group

SUMMARY:
This quasi-experimental two-group pretest-posttest study examined the effects of an interpersonal communication skills training program on medication adherence in patients with schizophrenia, measured at pre-intervention, post-intervention, and one-month follow-up.

Research Hypotheses

1. The experimental group receiving the interpersonal communication skills training program will show higher mean treatment adherence scores post-intervention and at one-month follow-up compared to baseline.
2. The experimental group will show higher mean treatment adherence scores post-intervention and at one-month follow-up than the control group receiving routine nursing care.

DETAILED DESCRIPTION:
Intervention : Interpersonal Communication Skills Training Program This program was developed based on DeVito's communication theory and integrated with the positive reinforcement-based interpersonal communication training developed by Thiengwiriyakul et al.(11) The program comprises six sessions: 1) Positive Communication 2) Equal Communication 3) Empathic Communication 4) Supportive Communication 5) Open Communication and 6) Relationship-Building Communication. The intervention was conducted three times per week, 60 minutes per session, over a two-week period.

Usual Care :

Usual care is defined as the provision of standard psychiatric nursing interventions consistent with usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 20-59 with an ICD-10 schizophrenia diagnosis(F20.0-F20.9).
2. History of psychiatric readmission due to medication non-adherence
3. Mild psychiatric symptoms(Thai BPRS score ≤ 36).
4. Poor interpersonal communication skills(score ≤ 1.50 on Thiengviriya et al.'s assessment tool
5. Low to moderate medication adherence(score ≤ 42 on Uthaiphan & Daengdomyut's scale
6. Able to read, write, speak, and without hearing/visual impairments.
7. Had a primary caregiver post-discharge.
8. Provided informed consent voluntarily.

Exclusion Criteria:

Patients with other psychiatric comorbidities(e.g., depression, bipolar disorder, anxiety, or substance-induced psychosis)

Ages: 20 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Behavior | Before the intervention, Immediately after the intervention , 1 month follow-up
  Treatment adherence refers to the extent to which patients with schizophrenia follow their prescribed medication regimen, assessed using the 16-item Treatment Adherence Behavior Assessment Scale (Uthaipan & Daengdomyut, 2013) It has been validated for content with a content validity index (CVI) of 0.88 and demonstrates good reliability with a Cronbach's alpha of 0.85. It consists of 16 items rated on a 4-point Likert scale (Always, Often, Occasionally, Never), divided into two parts: 1) Items 1-8: behaviors related to medication adherence. 2) Items 9-16: abilities to recognize and manage side effects. Seven items are negatively worded (Items 1, 2, 3, 7, 8, 12, 15), and nine items are positively worded (Items 4, 5, 6, 9, 10, 11, 13, 14, 16). The scoring is interpreted as follows: 1) ≤ 21 points: Low adherence 2) 21-42 points: Moderate adherence 3) ≥ 43 points: High adherence

CONTACTS AND LOCATIONS:
Overall Officials: Arunee Roongrusamee, Dip.N.S., Study Chair — Prasrimahabhodi Psychiatric Hospital, Ubon Ratchathani, 34000, Thailand; Palida Phalasak, M.N.S, Principal Investigator — Prasrimahabhodi Psychiatric Hospital, Ubon Ratchathani, 34000, Thailand; Aungkhana Chaiyarak, Dip.N.S., Principal Investigator — Prasrimahabhodi Psychiatric Hospital, Ubon Ratchathani, 34000, Thailand; Sakda Khumkom, Ph.D., Principal Investigator — Institute of Nursing, Suranaree University of Technology, Nakhon Ratchasima, 30000, Thailand; Thanakamon Leesri, Ph.D., Principal Investigator — Institute of Nursing, Suranaree University of Technology, Nakhon Ratchasima, 30000, Thailand
Locations (1):
- Prasrimahabhodi Psychiatric Hospital, ,Thailand, Nai Muang, Changwat Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Statement:
  Individual participant data (IPD) will be made available following publication of the research article and will remain accessible for 10 years thereafter.
Supporting Information: Study Protocol
Time Frame: 10 years thereafter.
Access Criteria: Access instructions will be provided at that time

REFERENCES:
- [Result] He H, Liu Q, Li N, Guo L, Gao F, Bai L, Gao F, Lyu J. Trends in the incidence and DALYs of schizophrenia at the global, regional and national levels: results from the Global Burden of Disease Study 2017. Epidemiol Psychiatr Sci. 2020 Jan 13;29:e91. doi: 10.1017/S2045796019000891. PMID 31928566
- [Result] Charlson FJ, Ferrari AJ, Santomauro DF, Diminic S, Stockings E, Scott JG, McGrath JJ, Whiteford HA. Global Epidemiology and Burden of Schizophrenia: Findings From the Global Burden of Disease Study 2016. Schizophr Bull. 2018 Oct 17;44(6):1195-1203. doi: 10.1093/schbul/sby058. PMID 29762765
- [Result] Semahegn A, Torpey K, Manu A, Assefa N, Tesfaye G, Ankomah A. Psychotropic medication non-adherence and its associated factors among patients with major psychiatric disorders: a systematic review and meta-analysis. Syst Rev. 2020 Jan 16;9(1):17. doi: 10.1186/s13643-020-1274-3. PMID 31948489
- [Result] While A. Medication adherence: understanding the issues and finding solutions. Br J Community Nurs. 2020 Oct 2;25(10):474-479. doi: 10.12968/bjcn.2020.25.10.474. PMID 33030359
- [Result] Tan XH, Foo MA, Lim SLH, Lim MBXY, Chin AMC, Zhou J, Chiam M, Krishna LKR. Teaching and assessing communication skills in the postgraduate medical setting: a systematic scoping review. BMC Med Educ. 2021 Sep 9;21(1):483. doi: 10.1186/s12909-021-02892-5. PMID 34503497
- [Result] Riedl L, Nagels A, Sammer G, Straube B. A Multimodal Speech-Gesture Training Intervention for Patients With Schizophrenia and Its Neural Underpinnings - the Study Protocol of a Randomized Controlled Pilot Trial. Front Psychiatry. 2020 Mar 6;11:110. doi: 10.3389/fpsyt.2020.00110. eCollection 2020. PMID 32210849
- [Result] Combs DR, Adams SD, Penn DL, Roberts D, Tiegreen J, Stem P. Social Cognition and Interaction Training (SCIT) for inpatients with schizophrenia spectrum disorders: preliminary findings. Schizophr Res. 2007 Mar;91(1-3):112-6. doi: 10.1016/j.schres.2006.12.010. Epub 2007 Feb 12. PMID 17293083
- [Result] Park Y, Han K. Development and evaluation of a Communication Enhancement Program for People with Chronic Schizophrenia: A quasi-experimental pretest-posttest design study. Appl Nurs Res. 2018 Aug;42:1-8. doi: 10.1016/j.apnr.2018.04.007. Epub 2018 Apr 25. PMID 30029708
- [Result] Maassen E, Buttner M, Brocker AL, Stuke F, Bayer S, Hadzibegovic J, Just SA, Bertram G, Rau R, von Haebler D, Lempa G, Montag C. Measuring Emotional Awareness in Patients With Schizophrenia and Schizoaffective Disorders. Front Psychol. 2021 Nov 11;12:725787. doi: 10.3389/fpsyg.2021.725787. eCollection 2021. PMID 34858263
- [Result] Uzun G, Lok N. Effect of emotional awareness skills training on emotional awareness and communication skills in patients with schizophrenia: A Randomized Controlled Trial. Arch Psychiatr Nurs. 2022 Jun;38:14-20. doi: 10.1016/j.apnu.2022.01.005. Epub 2022 Jan 22. PMID 35461642
- See also: fact- sheets of schizophrenia from WHO — http://www.who.int/news-room/fact-sheets/detail/schizophrenia